CLINICAL TRIAL: NCT06881381
Title: Investigation of Swallowing Complaints and Oral Sensory Problems in Children with a History of Preterm Birth
Brief Title: Swallowing and Oral Sensory Complaints in Preterm Children
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Hilal Berber Çiftci, PhD, Medipol University
Other Study IDs: MEAH
Record Dates: First submitted 2025-03-06; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Prematurity; Dysphagia; Feeding Disorder of Infancy or Early Childhood
MeSH Terms: conditions — Premature Birth; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Inclusion criteria were having a preterm child

SUMMARY:
Objective Preterm children face an elevated risk of neurodevelopmental delays and feeding difficulties, necessitating early assessment to support their long-term health. This study investigates swallowing disorders and oral sensory problems in children aged 3-10 years born preterm.

Methods Parents of preterm children completed two validated tools: the Pediatric Eating Assessment Tool (PEDI-EAT-10) to assess swallowing difficulties and the Oral Sensory Profile (Oral-SP) to evaluate oral sensory processing. Data collected included age, gender, gestational age, height, weight, neonatal intensive care unit (NICU) stay duration, feeding methods (e.g., tube feeding, pacifier, bottle use), medical history, and prior interventions like speech-language therapy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were having a preterm child (born before 37 weeks), aged 3-10 years, being Turkish-speaking, and volunteering.

Exclusion Criteria:

Participants were excluded if they withdrew during data collection.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants were parents of children attending a state hospital's Pediatric Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2024-11-24 (Actual)

PRIMARY OUTCOMES:
gestational age | 24-37 week

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the corresponding author. The data are not publicly available due to restrictions their containing information that could compromise the privacy of research participants.

REFERENCES:
- [Background] Cerro N, Zeunert S, Simmer KN, Daniels LA. Eating behaviour of children 1.5-3.5 years born preterm: parents' perceptions. J Paediatr Child Health. 2002 Feb;38(1):72-8. doi: 10.1046/j.1440-1754.2002.00728.x. PMID 11869405
- See also: Ministry of Health. Premature birth statistics. — https://dosyasb.saglik.gov.tr/Eklenti/48055/0/siy2022eng050420241pdf.pdf
- Available data/document: Study Protocol — https://docs.google.com/document/d/19ZwAv6y0UUaSa_Hjb3jlzuhMfTro0Y6p/edit?usp=drive_link&ouid=101334879348395838064&rtpof=true&sd=true — STUDY PROTOKOL DIAGRAM